CLINICAL TRIAL: NCT02999867
Title: Effect of Triticale, Mung Bean and Adzuki Bean Intervention on Metabolic and Nutritional Status of Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Triticale, Mung Bean and Adzuki Bean Intervention on Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PUMCH-ZS-1048
Record Dates: First submitted 2016-12-07; First posted 2016-12-21 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2017-08

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — subtilisin inhibitor, Vigna angularis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M1 triticale and mung bean (Experimental): M1: triticale and mung bean as a processed food is assigned to patients at a dose of 50-100 g/d for 30-day dietary intervention.
  Interventions: Dietary Supplement: triticale and mung bean
- M2 adzuki bean (Experimental): M2: adzuki bean as a processed food is assigned to patients at a dose of 50-100 g/d for 30-day dietary intervention.
  Interventions: Dietary Supplement: adzuki bean

INTERVENTIONS:
Dietary Supplement: triticale and mung bean — subjects are assigned to intake of triticale and mung bean for 30 days
  Other Names: M1 triticale and mung bean
  Arms: M1 triticale and mung bean
Dietary Supplement: adzuki bean — subjects are assigned to intake of adzuki bean for 30 days
  Other Names: M2 adzuki bean
  Arms: M2 adzuki bean

SUMMARY:
This study is designed to evaluate short term effect of triticale, mung bean and adzuki bean intervention for health improvement in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The study will evaluate the effect of triticale, mung bean and adzuki bean on metabolic and nutritional status of patients with type 2 diabetes after 30 days of intervention. Patients will be assigned to control or intervention group (A diet including triticale and mung bean; B diet including adzuki bean). Blood and urine samples will be collected at baseline and after 30 days of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 30 and 65 years
2. patients has been diagnosed as type 2 diabetes mellitus
3. Patients who like to be followed up for 2 months.

Exclusion Criteria:

1. Women in pregnancy or lactation.
2. Individuals with a history of severe kidney disease, cardiovascular disease, stroke, cancer, or psychological disorders.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
response to the dietary intervention by the change from baseline in blood glucose at 30-day | baseline and 30 d
response to the dietary intervention by the change from baseline in lipid profile at 30-day | baseline and 30 d
response to the dietary intervention by the change from baseline in insulin resistance at 30-day | baseline and 30 d

SECONDARY OUTCOMES:
response to the dietary intervention by the change from baseline in renal function at 30-day | baseline and 30 d
response to the dietary intervention by the change from baseline in liver function at 30-day | baseline and 30 d
response to the dietary intervention by the change from baseline in inflammation result at 30-day | baseline and 30 d
response to the dietary intervention by the change from baseline in folic acid absorption at 30-day | baseline and 30 d
response to the dietary intervention by the change from baseline in iron absorption at 30-day | baseline and 30 d

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Liu, master, Study Director — Department of Nutrition, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided